CLINICAL TRIAL: NCT02419950
Title: Impact of Mesh Fixation on Chronic Pain in Total Extraperitoneal (TEP) Inguinal Hernia Repair - a National Register Based Study
Brief Title: Mesh Fixation inTEP Inguinal Hernia Repair
Acronym: register
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Agneta Montgomery, PhD, MD, Skane University Hospital
Other Study IDs: 634/2008
Record Dates: First submitted 2014-09-24; First posted 2015-04-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; TEP; chronic pain; male sex; mesh fixation; quality of life; national register
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No fixation of mesh in TEP: Patient having no mechanical fixation of the mesh in TEP. This will include both no fixation at all och glue fixation of the mesh in total extraperitoneal placement of mesh by endoscopic technique
  Interventions: Device: Fixation of mesh in TEP
- Fixation of mesh in TEP: Patients having fixation of the mesh using mechanical, non absorbable fixating devices.This will include mechanical fixation of the mesh in total extraperitoneal placement of mesh by endoscopic technique
  Interventions: Device: Fixation of mesh in TEP

INTERVENTIONS:
Device: Fixation of mesh in TEP — An endoscopic operative technique were mesh for preperitonelal placement in patients with inguinal hernias can be fixated in Place or left without fixation
  Other Names: Total Extraperitoneal Patch

SUMMARY:
Mesh fixation is used to prevent recurrence in TEP to the potential cost of pain. The aim was to evaluate the impact of permanent fixation (PF) versus non-permanent fixation (N-PF) of mesh in TEP repair for a primary inguinal hernia regarding chronic pain. A cohort of patients were studied for pain interfering with sexual activety. The hyopthesis is that fixation causes pain.

DETAILED DESCRIPTION:
Mesh fixation is used to prevent recurrence in TEP to the potential cost of pain. The aim was to evaluate the impact of permanent fixation (PF) versus non-permanent fixation (N-PF) of mesh in TEP repair for a primary inguinal hernia regarding chronic pain.

Men between 30 and 75 years, consecutively registered in Swedish Hernia Register (SHR) for a TEP repair between 2005 and 2009 were included. A questionnaire was sent in 2010 including a general questionnaire, SF-36 and Inguinal Pain Questionnaire (IPQ). Primary endpoint was question two in IPQ, "worst pain you felt in the operated groin during this past week". Pain was defined as "pain present that could not be ignored". In adition a specific questionnair developed by the research group on pain and problems during sexual activiety were sent to patients between 30-60 years of age.

The register was checked for long term recurrent operations.

ELIGIBILITY:
Inclusion Criteria:

* Male between 30-75 years.
* Primary inguinal hernia

Exclusion Criteria:

* Emergency operation
* Operated for recurrence
* Deaths

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men between 30-75 years with primary inguinal hernia
Sampling Method: Non-Probability Sample
Enrollment: 1110 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Chronic pain | 5 years
  Chronic pain is meassured using an Enquirer sent to the patients by mail containing general questions to be able to exclude patients having a chronic pain problem due to other causes than the hernia (like back pain and other operations in the area) SF 36 questionnair for global measures of physical and mental Health and an validated inguinal hernia specific questionnaire for measuring pain, IPQ (Inguinal Pain Questionnair) was used

SECONDARY OUTCOMES:
Sexual problems due to inguinal pain problems after hernia surgery | 2-5 years
  A specific questionnair, localy developed, for deltaled information on type, frequency, duration,intensety, disabeling and location of pain together with questions on interferance with errection, ejacculation as well as interferance with general well beeing.
A second operation for a recurrence | 5-7 years
  Measured as a reoperation reported in the national register

CONTACTS AND LOCATIONS:
Overall Officials: Agneta Montgomery, MD, PhD, Principal Investigator — University of Lund, Sweden
Locations (1):
- University of Lund,, Malmo, Sweden

REFERENCES:
- [Background] Franneby U, Gunnarsson U, Andersson M, Heuman R, Nordin P, Nyren O, Sandblom G. Validation of an Inguinal Pain Questionnaire for assessment of chronic pain after groin hernia repair. Br J Surg. 2008 Apr;95(4):488-93. doi: 10.1002/bjs.6014. PMID 18161900
- [Background] Kehlet H, Bay-Nielsen M, Kingsnorth A. Chronic postherniorrhaphy pain--a call for uniform assessment. Hernia. 2002 Dec;6(4):178-81. doi: 10.1007/s10029-002-0082-0. Epub 2002 Sep 20. PMID 12424597
- [Background] Eklund A, Rudberg C, Smedberg S, Enander LK, Leijonmarck CE, Osterberg J, Montgomery A. Short-term results of a randomized clinical trial comparing Lichtenstein open repair with totally extraperitoneal laparoscopic inguinal hernia repair. Br J Surg. 2006 Sep;93(9):1060-8. doi: 10.1002/bjs.5405. PMID 16862612
- [Background] Aasvang EK, Mohl B, Bay-Nielsen M, Kehlet H. Pain related sexual dysfunction after inguinal herniorrhaphy. Pain. 2006 Jun;122(3):258-263. doi: 10.1016/j.pain.2006.01.035. Epub 2006 Mar 20. PMID 16545910
- [Background] Kaul A, Hutfless S, Le H, Hamed SA, Tymitz K, Nguyen H, Marohn MR. Staple versus fibrin glue fixation in laparoscopic total extraperitoneal repair of inguinal hernia: a systematic review and meta-analysis. Surg Endosc. 2012 May;26(5):1269-78. doi: 10.1007/s00464-011-2025-2. Epub 2012 Feb 21. PMID 22350225